CLINICAL TRIAL: NCT04098302
Title: Dutasteride Treatment for Reducing Heavy Drinking in AUD: Predictors of Efficacy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Covault, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-147-2; P50AA027055 (NIH)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Dutasteride

STUDY DESIGN:
Intervention Model Description: The study consists of two 12-week phases, the first being a 12-week parallel-groups comparison of dutasteride and placebo to evaluate the safety and efficacy of dutasteride 1 mg/day in reducing the likelihood of drinking and heavy drinking in treatment-seeking men and women with alcohol use disorder. In the second 12-week phase, responders in phase 1 (defined as a ≥60% reduction in SD/wk for weeks 9-12 compared with screening) will continue on their initial medication assignment, while non-responder subjects treated with placebo in phase 1 will be given dutasteride during phase 2, and non-responder subjects treated with dutasteride in phase 1 will receive naltrexone daily in phase 2. This design maintains double blind conditions in both phases 1 and 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: UConn Health Investigational Pharmacy will randomize to dutasteride vs. placebo for phase 1 at baseline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dutasteride (Active Comparator): two 0.5 mg capsules of dutasteride daily
  Interventions: Drug: Dutasteride Capsules
- placebo capsule (Placebo Comparator): inactive placebo matched in appearance with dutasteride capsules
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: Dutasteride Capsules — 1 mg/day oral dutasteride (2 x 0.5 mg capsules)
  Other Names: Avodart
  Arms: dutasteride
Drug: Placebo Capsules — Placebo capsules with matching appearance as Dutasteride Capsules
  Other Names: inactive placebo
  Arms: placebo capsule

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of dutasteride in reducing drinking and heavy drinking in men and women with alcohol use disorder. The investigators hypothesize that dutasteride 1 mg per day will be well tolerated in this patient population and that, compared to placebo treatment, dutasteride will result in a greater reduction in drinks per week and in the frequency of heavy drinking days.

DETAILED DESCRIPTION:
Heavy drinking remains a significant public health problem and is frequently under treated. Although several medications have been shown to help patients stop or reduce drinking, additional medication options are needed as there is considerable variability in effectiveness or tolerability of existing medications for individual patients. Additionally, identification of individual subject level predictors of efficacy are needed to better personalize pharmacotherapy treatment recommendations. This study will seek to replicate and extend our results showing efficacy of a novel medication dutasteride for reducing drinking and will examine potential easily measured predictors of response.

Dutasteride is a widely prescribed medication for benign prostatic hypertrophy and androgenic hair loss that also modulates the elimination of cortisol and the production of some neuroactive steroids. Changes in the regulation of cortisol and neuroactive steroids have each been suggested as factors which may contribute to the maintenance of alcohol dependence. Data from a recently completed first randomized placebo controlled trial of dutasteride for AUD in a sample of male drinkers, indicates that dutasteride is well tolerated in alcoholics and has efficacy in helping subjects reduce drinking. Additionally, results indicate that dutasteride may be particularly helpful for patients who drink to cope with anxiety and negative emotions, a group of patients with poor response to other treatments.

This 24-week treatment study will use an innovative randomized placebo controlled step therapy design to examine the safety and efficacy of dutasteride to reduce drinking by treatment seeking women and men with hazardous levels of alcohol use. At 12-weeks placebo non-responders will transition to dutasteride and dutasteride non-responders will transition to naltrexone, an FDA approved medication with demonstrated efficacy for reducing heavy drinking. 12-week responders (reduction in drinks/week of 60% or greater compared with screening) will continue for an additional 12-weeks on their initial study medication assignment (dutasteride or placebo).

Additionally, the investigators will examine several baseline measures as predictors of dutasteride efficacy, including drinking to cope, anxiety, adverse child events, and perceived life stress as well as stress resilient vs. reactive genotypes of FKBP5 a chaperone protein involved in regulation of glucocorticoid, androgen and progesterone receptor function.

ELIGIBILITY:
Inclusion Criteria:

* men and women age 35 to 70 yo inclusive
* have an average weekly ethanol consumption of >24 SD for men and >18 for women and at least 2 HDD/wk over the 8 weeks prior to screening
* current DSM-5 AUD
* no evidence of significant cognitive impairment
* for women of child-bearing potential (i.e., no hysterectomy, bilateral oophorectomy, or tubal ligation; or <2 years postmenopausal) must be non-lactating, practicing a reliable method of birth control and agree to continue such throughout the study and for 6 months following participation, and have a negative serum pregnancy test prior to initiation of treatment.

Exclusion Criteria:

* history of serious alcohol withdrawal symptoms (e.g., perceptual distortions, seizures, delirium, or hallucinations)
* subjects who on clinical examination by a physician are deemed to be too severely alcohol dependent to permit them to participate in a pbo-controlled study (e.g., evidence of serious adverse medical or psychiatric effects that are exacerbated by heavy drinking and would, for safety reasons, lead the physician to urge the patient to be totally abstinent and engage in an empirically supported treatment)
* current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation, including direct bilirubin more than 2.5 times the upper limit of normal or transaminase elevations 5 times the upper limit of normal (the investigators will not exclude patients with hypertension, diabetes, asthma or other common medical conditions, if these are adequately controlled and the patient has an ongoing relationship with a primary care provider)
* have a serious psychiatric illness on the basis of history or psychiatric examination (i.e., schizophrenia, active clinically significant mood episode of bipolar disorder or major depression, organic mental disorder, current clinically significant eating disorder, or substantial suicide or violence risk)
* have a current DSM-5 diagnosis of moderate drug use disorder (other than caffeine or nicotine dependence)
* currently taking finasteride, dutasteride, medication for treatment of AUD, or chronic use of opioid pain medication
* are considered by the investigators to be an unsuitable candidate for an investigational drug

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Covault, MD, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Via postings at UConn Health and radio advertisements
Pre-assignment Details: Of the 180 consented, 10 were screen failures and 3 withdrew after screening visit. Five participants did not attend baseline visit to receive medication and 7 did return after baseline visit leaving 155 as the phase 1 modified intention to treat sample (75 dutasteride arm and 80 placebo arm).
Groups:
- Dutasteride - Naltrexone: Phase 1 (week 1-12) dutasteride arm participants with <60% reduction in drinks per week assigned to naltrexone 50 mg daily for Phase 2 (weeks 13-24)
- Placebo - Dutasteride: Phase 1 (week 1-12) placebo arm participants with <60% reduction in drinks per week assigned to dutasteride 1mg daily for Phase 2 (weeks 13-24)
Period: Wk 1-12 Phase 1 Dutasteride or Placebo
Arm/Group | Dutasteride | Placebo Capsule | Dutasteride - Naltrexone | Placebo - Dutasteride
Started | 75 | 80 | 0 | 0
Completed | 65 | 66 | 0 | 0
Not Completed | 10 | 14 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 11 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 0 | 0
Period: Wk 13-24 for Phase 1 Non-responders
Arm/Group | Dutasteride | Placebo Capsule | Dutasteride - Naltrexone | Placebo - Dutasteride
Started | 0 | 0 | 49 | 59
Completed | 0 | 0 | 44 | 53
Not Completed | 0 | 0 | 5 | 6
Not completed — Lost to Follow-up | 0 | 0 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dutasteride: two 0.5 mg capsules of dutasteride daily for 12 weeks
- Placebo Capsule: inactive placebo matched in appearance with dutasteride capsules daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Dutasteride | Placebo Capsule | Total
Number analyzed (Participants) | 75 | 80 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (9.3) | 55.5 (8.9) | 56.3 (91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 40 | 48 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 68 | 79 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 74 | 77 | 151
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 75 | 80 | 155
Number of heavy drinking days per week [Mean (Standard Deviation); unit: Heavy drinking days per week] — number of heavy drinking days (four or more drinks in a day for women and five or more drinks in a day for men) per week
  Heavy drinking days per week | 5.4 (1.8) | 5.6 (1.7) | 5.5 (1.7)
Drinks per week [Mean (Standard Deviation); unit: drinks per week] — number of standard drinks per week (14 gr alcohol)
  drinks per week | 43.2 (21.9) | 43.5 (18.5) | 43.4 (20.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Heavy Drinking Days Per Week for Dutasteride vs. Placebo Groups
Description: The number of heavy drinking days per week (i.e., four or more drinks in a day for women and five or more drinks in a day for men). The values listed in outcome table are the average HDD per week for the last 4 weeks (9-12) of phase 1 treatment. The generalized linear mixed model analysis considered all data from the ITT sample (75 dutasteride and 80 placebo participants)
Time Frame: 12 weeks (from initiation to end of treatment phase 1)
Population: Participants who attended and provided outcome data for at least one study visit following baseline session.
Measure: Mean (Standard Error); unit: Heavy Drinking Days per week
Arm/Group | Dutasteride | Placebo Capsule
Number analyzed (Participants) | 75 | 80
Heavy Drinking Days per week | -2.24 (0.33) | -1.41 (0.28)
Statistical Analysis 1: Comparison: Dutasteride vs Placebo Capsule; Test type: Superiority; p = 0.012, Mixed Models Analysis

2. Primary Outcome: Change in Drinks Per Week in Dutasteride vs. Placebo Groups
Description: Change in the number of drinks per week during treatment phase 1 of study (week 1-12). The values listed in the outcome table are the average drinks per week for the last 4 weeks of treatment (week 9-12). The generalized linear mixed model analysis considered all data from the ITT sample (75 dutasteride and 80 placebo participants)
Time Frame: 12 weeks (from initiation to end of treatment phase 1)
Population: Participants who attended and provided outcome data for at least one study visit following baseline session.
Measure: Mean (Standard Error); unit: Drinks per week
Arm/Group | Dutasteride | Placebo Capsule
Number analyzed (Participants) | 75 | 80
Drinks per week | -14.16 (2.49) | -7.72 (2.16)
Statistical Analysis 1: Comparison: Dutasteride vs Placebo Capsule; Test type: Superiority; p = 0.019, Mixed Models Analysis

3. Other Pre Specified Outcome: Change in Heavy Drinking Days Per Week for Phase 2 Naltrexone vs Dutasteride Groups
Description: The number of heavy drinking days per week (i.e., four or more drinks in a day for women and five or more drinks in a day for men) for phase 1 non-responders (<60% reduction in drinks per week) during phase 2 comparing naltrexone 50 mg and dutasteride 1 mg daily. The values listed in outcome table are the mean change in HDD per week for the last 4 weeks (wk 21-24) of phase 2 relative to drinking at beginning of phase 2 treatment. treatment.
Time Frame: 12 weeks (week 13 to end of treatment phase 2, week 24)
Population: Phase 2 (wk13-24) completers. The generalized linear mixed model analysis considered all data from the phase 2 ITT sample (phase 1 non-responders with <60% reduction in drinks per week (49 phase 1 dutasteride-phase 2 naltrexone and 59 phase 1 placebo-phase 2 dutasteride participants).
Measure: Mean (Standard Error); unit: Heavy drinking days per week
Arm/Group | Dutasteride - Naltrexone | Placebo - Dutasteride
Number analyzed (Participants) | 44 | 53
Heavy drinking days per week | -1.45 (0.26) | -0.54 (0.25)
Statistical Analysis 1: Comparison: Dutasteride - Naltrexone vs Placebo - Dutasteride; Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Other Pre Specified Outcome: Change in Drinks Per Week in Phase 2 Naltrexone vs. Dutasteride Groups
Description: The number of drinks per week for phase 1 non-responders (<60% reduction in drinks per week) during phase 2 comparing naltrexone 50 mg and dutasteride 1 mg daily. The values listed in outcome table are the mean change in drinks per week for the last 4 weeks (wk 21-24) relative to drinking at beginning of phase 2 treatment.
Time Frame: 12 weeks (week 13 to end of treatment phase 2, week 24)
Population: Phase 2 completers (wk 13-24). The generalized linear mixed model analysis considered all data from the phase 2 ITT sample (phase 1 non-responders. 49 phase 1 dutasteride-phase 2 naltrexone and 59 phase 1 placebo-phase 2 dutasteride participants).
Measure: Mean (Standard Error); unit: drinks per week
Arm/Group | Dutasteride - Naltrexone | Placebo - Dutasteride
Number analyzed (Participants) | 44 | 53
drinks per week | -7.29 (1.37) | -5.31 (1.48)
Statistical Analysis 1: Comparison: Dutasteride - Naltrexone vs Placebo - Dutasteride; Test type: Superiority; p = 0.29, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Phase 1 first 12 weeks: dutasteride vs. placebo arms data collected at bi-weekly visits (week 2 to week 12) Phase 2 second 12 weeks for phase 1 participants with <60% reduction drinks per week transition to either dutasteride or naltrexone: placebo-dutasteride vs. dutasteride-naltrexone arms data collected at bi-weekly Phase 2 visits (week 14 to week 24)
Description: Participants provided subjective reports of adverse events at each bi-weekly study visit using the Systematic Assessment for Treatment Emergent Effects (SAFTEE) interview, a widely used tool for systematic assessment of adverse events.
Groups:
- Placebo Capsule: inactive placebo matched in appearance with dutasteride capsules for 12 weeks
Arm/Group | Dutasteride | Placebo Capsule | Dutasteride - Naltrexone | Placebo - Dutasteride
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/80 | 0/49 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/80 | 0/49 | 2/59
Other Adverse Events (participants affected / at risk) | 46/75 | 41/80 | 34/49 | 33/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride (N=75) | Placebo Capsule (N=80) | Dutasteride - Naltrexone (N=49) | Placebo - Dutasteride (N=59)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — subject reported history of pancreatitis was admitted to local hospital for acute pancreatitis at study week 18. subject had treatment with placebo week1-12 and then dutasteride 1 mg daily week 13-18 and continued to drink alcohol.
fall from step ladder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject presented to emergency department after fall from step ladder at home while sober at study week 19. Rib fracture identified and discharged home. Subject received daily placebo wk 1-12 and then dutasteride 1mg daily wk 13-24.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dutasteride (N=75) | Placebo Capsule (N=80) | Dutasteride - Naltrexone (N=49) | Placebo - Dutasteride (N=59)
Nausea (Gastrointestinal disorders) | 8 (18) | 5 (8) | 11 (20) | 6 (12)
Muscle or body ache (Musculoskeletal and connective tissue disorders) | 8 (10) | 7 (8) | 9 (33) | 2 (8)
Itching (Skin and subcutaneous tissue disorders) | 7 (12) | 4 (6) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 6 (12) | 3 (4) | 4 (13) | 3 (13)
Dizzy or lightheaded (General disorders) | 6 (8) | 6 (10) | 4 (4) | 4 (9)
Numbness or Tingling around Mouth, Fingers, or Toes (Nervous system disorders) | 6 (9) | 6 (17) | 1 (1) | 2 (6)
Decreased libido (Reproductive system and breast disorders) | 5 (21) | 3 (5) | 1 (3) | 2 (9)
Irritability (Psychiatric disorders) | 5 (11) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (7) | 5 (10) | 5 (10) | 3 (7)
Difficulty sleeping (Nervous system disorders) | 4 (7) | 2 (7) | 5 (13) | 9 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT04098302/Prot_SAP_001.pdf